CLINICAL TRIAL: NCT01993927
Title: Voglibose Tablets 0.2 / Voglibose Oral Disintegrant (OD) Tablets 0.2 Special Drug Use Surveillance "Long-term Use in Patients With Impaired Glucose Tolerance"
Brief Title: Voglibose Tablets 0.2 / OD Tablets 0.2 Special Drug Use Surveillance "Long-term Use in Patients With Impaired Glucose Tolerance"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 340-012; JapicCTI-132304 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Impaired Glucose Tolerance
Keywords: Drug Therapy
MeSH Terms: conditions — Glucose Intolerance | interventions — voglibose; AO 128

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Voglibose 0.2 mg or OD Tablets 0.2 mg: Voglibose 0.2 mg or OD Tablets 0.2 mg will be administered orally three times daily immediately before each meal.
  Interventions: Drug: Voglibose

INTERVENTIONS:
Drug: Voglibose — Voglibose Tablets / Voglibose OD Tablets
  Other Names: Basen Tablets, AO-128

SUMMARY:
The purpose of this study is to determine the safety and efficacy of long-term use of Voglibose (Basen) to prevent progression to type 2 diabetes mellitus in participants with impaired glucose tolerance in the routine clinical setting.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of Voglibose (Basen) designed to determine the safety and efficacy of long-term use of Voglibose (Basen) to prevent progression to type 2 diabetes mellitus in participants with impaired glucose tolerance in the routine clinical setting.

Particioants will be patients with impaired glucose tolerance. The planned sample size is 1,000.

The usual adult dosage is 0.2 mg of voglibose administered orally three times daily immediately before each meal.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria ([1] to [3]) to be included in this study:

  1. Determined as having IGT (defined as fasting blood glucose < 126 mg/dL and 2-hour post 75-g oral glucose tolerance test [OGTT] blood glucose of 140-199 mg/dL) without improvement despite treatment with diet therapy and exercise therapy for 3-6 months
  2. Meets any of the following conditions:

     (i) Concurrently has hypertension*1 (ii) Concurrently has dyslipidemia*2 (iii) Is obese (BMI ≥25 kg/m^2) (iv) Has a family history of diabetes mellitus in relatives to the second degree as defined by Japanese law*3
  3. Regularly visits the study site and can be observed for 72 weeks

     * 1: Hypertension: Patients with systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, or patients on oral antihypertensive medication.
     * 2: Dyslipidaemia: Participants with any of the following conditions or participants on oral antidyslipidemic medication
* Hyper LDL cholesterolemia (fasting LDL-cholesterol ≥140 mg/dL)
* Hypo HDL cholesterolemia (fasting HDL-cholesterol < 40 mg/dL)
* Hypertriglyceridemia (fasting triglyceride ≥150 mg/dL) *3: Relatives to the second degree of consanguinity refer to blood relatives who are the subject's "father or mother, grandfather or grandmother, brothers or sisters, children, or grandchildren." Note that these do not include spouse's relatives.

Exclusion Criteria:

* Participants meeting either of the following criteria ([1] or [2]) will be excluded:

  1. Previously diagnosed with diabetes mellitus
  2. Has any contraindications to Basen as specified below:

     (i) Severe ketosis, diabetic coma or precoma (ii) Severe infection, perioperative state, or serious trauma (iii) History of hypersensitivity to any ingredients of Basen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with impaired glucose tolerance
Sampling Method: Non-Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 130 investigative sites in Japan, from 18-November-2009 to 31-August-2013.
Pre-assignment Details: Participants, who had determined as having impaired glucose tolerance (IGT) without improvement despite treatment with diet therapy and exercise therapy for 3-6 months, were enrolled to receive voglibose 0.2 milligram (mg) orally, three times daily, up to 72 months (approximately 1 year and 6 months).
Groups:
- Voglibose 0.2 mg or OD Tablets 0.2 mg: Voglibose 0.2 mg or OD Tablets 0.2 mg was administered orally three times daily immediately before each meal, up to 72 months (approximately 1 year and 6 months). Participants will receive interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Started | 742
Completed | 713
Not Completed | 29
Not completed — Case Report Forms Uncollected | 18
Not completed — Protocol Violation | 11

BASELINE CHARACTERISTICS:
Population: Safety/Efficacy Analysis Set was defined as all participants who were enrolled and completed the study. All data could be received as case report forms without major protocol violations.
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Number analyzed (Participants) | 713
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337
  Male | 376
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 713
Duration of Disease [Mean (Standard Deviation); unit: Months] — Mean Duration between start of study and first time of diagnosis of Impaired Glucose Tolerance (IGT) was reported.
  Months | 12.51 (23.708)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient (participants who were both outpatient and inpatient during some point at the time and 3 months prior to enrollment).
  Participants
    Outpatient | 706
    Inpatient | 2
    Inpatient and Outpatient | 5
Pregnancy Status [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    Not pregnant: number analyzed (Participants) | 337
    Not pregnant | 337
    Pregnant: number analyzed (Participants) | 337
    Pregnant | 0
History of Allergy [Count of Participants; unit: Participants]
  Had No History of Allergy | 623
  Had History of Allergy | 59
  Unknown | 31
Family History of Diabetes in Second-Degree Relatives [Count of Participants; unit: Participants]
  Had No Family History of Diabetes | 567
  Had Family History of Diabetes | 146
History of Obesity [Count of Participants; unit: Participants] — Number of Participants with 25 kg/m^2 or more as Body Mass Index were reported.
  Participants
    Had No History of Obesity | 410
    Had History of Obesity | 303
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 46
    Had Presence of Medical Complications | 667
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Presence of Medical History | 584
    Had Presence of Medical History | 126
    Unknown | 3
Height [Mean (Standard Deviation); unit: cm] | 160.21 (9.619)
Weight [Mean (Standard Deviation); unit: kg] | 63.21 (13.097)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 24.55 (3.873)
Drinking Habits [Count of Participants; unit: Participants]
  Never Drank | 404
  Ex-Drinker | 47
  Current Drinker | 261
  Unknown | 1
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 533
  Ex-Smoker | 87
  Current Smoker | 92
  Unknown | 1
Duration of Dietary and Exercise Therapies prior to the Administration of Voglibose [Count of Participants; unit: Participants]
  Not performed | 56
  < 3 months | 304
  ≥ 3 months < 6 months | 176
  ≥ 6 months < 1 year | 163
  ≥ 1 year | 14
Daily Activity Intensity Index [Count of Participants; unit: Participants] — Daily Activity Intensity Index is scored time in a day checked by investigators, assessing intensity of daily-life activities including five sub-scales which are Laying, Standing, Walking, Running and Exercising. Score range is from 1 (very mild activities in a day) to 4 (very strong activities in a day). Higher scores reflect stronger activities of participants in a day.
  Participants
    I (very mild activities in a day) | 159
    II (mild activities) | 302
    III (moderate/optimal) | 245
    IV (very strong activities in a day) | 7
75g OGTT Fasting Blood Glucose Level [Mean (Standard Deviation); unit: mg/dL] — OGTT; Oral glucose tolerance test. 75 g Oral glucose tolerance test measures blood glucose through blood samples drawn at 30, 60, 120 minutes following consumption of a 75 g glucose beverage.
  mg/dL | 105.3 (11.00)
75g OGTT Blood Glucose Level at 30 min after Dosing [Mean (Standard Deviation); unit: mg/dL] | 181.4 (28.45)
75g OGTT Blood Glucose Level at 2 hr after Dosing [Mean (Standard Deviation); unit: mg/dL] | 168.2 (17.42)
Fasting Blood Insulin Level [Mean (Standard Deviation); unit: mcU/mL] | 7.311 (4.8720)
Blood Insulin Level at 30 min after Dosing [Mean (Standard Deviation); unit: mcU/mL] | 38.122 (25.7354)
Blood Insulin Level at 2 hr after Dosing [Mean (Standard Deviation); unit: mcU/mL] | 69.405 (52.2083)
HbA1c (Japan DiabetesSociety; JDS Value) [Mean (Standard Deviation); unit: Percent] — HbA1c (JDS) shows a concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound. The 6.5% HbA1c is the JDS value, and is equivalent to the NGSP HbA1c value of 6.9%.
  Percent | 5.72 (0.399)
HbA1c (National Glycohemoglobin Standardization Program; NGSP Value) [Mean (Standard Deviation); unit: Percent] — HbA1c (NGSP) shows a concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound. The 6.5% HbA1c is the JDS value, and is equivalent to the NGSP HbA1c value of 6.9%.
  Percent | 6.11 (0.406)
Homeostasis Model Assessment of Insulin Resistance [Mean (Standard Deviation); unit: Percent score of insulin resistance] — Homeostasis Model assessment of insulin resistance measures insulin resistance, calculated by fasting insulin times fasting glucose, divided by a constant (405).
  Percent score of insulin resistance | 1.913 (1.3331)
Insulinogenic Index [Mean (Standard Deviation); unit: Score of insulinogenic Index] — Insulinogenic Index measures secretion of insulin, calculated by change from baseline in measured blood insulin at 30min (mcrU/ml), divided by change from baseline in measured blood glucose at 30min (mg/dl).
  Score of insulinogenic Index | 0.449 (0.3914)
Number of Risk Factor [Count of Participants; unit: Participants] — Reporting number of factors of risk which each participant had at study start. Factors included Glucose Intolerance, Complication of Hypertension, Complication of Hyperlipidemia, Obesity, Family History of Diabetes in Second-Degree Relatives
  Participants
    None | 0
    One Factor | 0
    Two Factors | 238
    Three Factors | 278
    Four Factors | 178
    Five Factors | 19
Compliance of Dietary Therapy at 6 Months prior to Study Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 187
  Compliance level of < 70% | 107
  Unknown | 419
Compliance of Dietary Therapy at 3 Months prior to Study Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 297
  Compliance level of < 70% | 212
  Unknown | 204
Compliance of Dietary Therapy at Treatment Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 391
  Compliance level of < 70% | 240
  Unknown | 82
Compliance of Exercise Therapy at 6 Months prior to Study Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 167
  Compliance level of < 70% | 120
  Unknown | 426
Compliance of Exercise Therapy at 3 Months prior to Study Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 260
  Compliance level of < 70% | 221
  Unknown | 232
Compliance of Exercise Therapy at Treatment Start [Count of Participants; unit: Participants]
  Compliance level of ≥ 70% | 331
  Compliance level of < 70% | 269
  Unknown | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Events
Time Frame: Up to Week 72
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Number analyzed (Participants) | 713
Participants | 88

2. Primary Outcome: Percentage of Participants With Progression to Type 2 Diabetes Mellitus (T2DM) During Treatment Period
Description: Percentage of participants who occurred progression of T2DM during treatment period was reported. Diagnostic criteria for progression of T2DM are: (1) "Blood glucose ≥200 mg/dL at any time, morning fasting blood glucose ≥126 mg/dL, or 2-hour post 75-g (Oral Glucose Tolerance Test) blood glucose ≥200 mg/dL. (2) Two or more glucose measurements obtained on different days that meet the above-mentioned criteria, or (3) A single glucose measurement meeting the above-mentioned criteria if the patient meets any of the following conditions: (i) Has typical symptoms of diabetes mellitus (e.g., dry mouth, polydipsia, polyuria, weight loss) (ii) HbA1C ≥6.5% (JDS value) (iii) Obvious diabetic retinopathy.
Time Frame: Up to Week 72
Population: Safety/Efficacy Analysis Set was defined as all participants who were enrolled and completed the study. Reported data was collected from received case report forms including the data, without major protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Number analyzed (Participants) | 708
Percentage of participants | 4.8

3. Secondary Outcome: Percentage of Participants With Normalization of Impaired Glucose Tolerance (IGT) During Treatment Period
Description: Percentage of participants who had normalization of Impaired Glucose Tolerance (IGT) during treatment period was reported. IGT normalization was determined by the survey physician based on the results of the 75-g oral glucose tolerance test (OGTT), glucose metabolism markers, and other data.
Time Frame: Up to Week 72
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Number analyzed (Participants) | 708
Percentage of participants | 11.3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Participants may be represented in more than 1 category.
Arm/Group | Voglibose 0.2 mg or OD Tablets 0.2 mg
Serious Adverse Events (participants affected / at risk) | 5/713
Other Adverse Events (participants affected / at risk) | 39/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voglibose 0.2 mg or OD Tablets 0.2 mg (N=713)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Eye disorders (Endocrine disorders) | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voglibose 0.2 mg or OD Tablets 0.2 mg (N=713)
Diarrhoea (Gastrointestinal disorders) | 14
Abdominal distension (Gastrointestinal disorders) | 14
Hepatic function abnormal (Hepatobiliary disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.